CLINICAL TRIAL: NCT07038252
Title: The Effect of Oral SPM Supplementation on INflammation-induced Vascular Ageing in Obese Hypertensive Patients
Acronym: SPIN-VA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other); The Company SOLUTEXGC, S.L (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP241105; 2025-A00108-41 (Other: French National Agency for the Safety of Medicines and Health Products (ANSM))
Record Dates: First submitted 2025-05-22; First posted 2025-06-26 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Obesity
MeSH Terms: conditions — Hypertension; Obesity | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm: active product is Oral SPM-enriched marine oil (Experimental): Active treatment product is Oral SPM-enriched marine oil (3 gr/day) 3 capsules after breakfast and 3 capsules after dinner, provided by Solutex.
  Interventions: Dietary Supplement: Oral SPM-enriched marine oil (LIPINOVA)
- Control arm :Placebo (olive oil) (Placebo Comparator): Placebo (olive oil) will be provided by Solutex too and will have the same appearance (3 capsules after breakfast and 3 capsules after dinner) as active
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral SPM-enriched marine oil (LIPINOVA) — LIPINOVA is an oral dietary supplement provided by Solutex, consisting of marine oil enriched in specialized pro-resolving mediator (SPM) precursors. Each daily dose (3 g/day) includes 1500 mg of omega-3 free fatty acids and a minimum of 520 mcg of SPM precursors (17-HDHA, 18-HEPE, 14-HDHA). The supplement is administered orally in 6 softgel capsules per day (3 after breakfast, 3 after dinner) over 12 weeks. It is used to investigate its effect on vascular function and inflammation in patients with obesity-related hypertension. The product is over-the-counter and commonly available in the EU, including France.
  Other Names: SPM-enriched marine oil; Omega-3 free fatty acids with SPM precursors; Specialized pro-resolving mediator supplement
  Arms: Experimental arm: active product is Oral SPM-enriched marine oil
Dietary Supplement: Placebo — Placebo capsules provided by Solutex, identical in appearance to LIPINOVA, contain refined olive oil with no active omega-3 fatty acids or SPM precursors. The placebo is administered orally in 6 softgel capsules per day (3 after breakfast, 3 after dinner) for 12 weeks, following a randomized, double-blind, crossover design. It serves as a control to evaluate the effects of SPM-enriched marine oil on vascular and inflammatory parameters in patients with obesity-related hypertension.
  Other Names: Olive oil capsules; Placebo SPM supplement
  Arms: Control arm :Placebo (olive oil)

SUMMARY:
Cardiovascular risk factors such as obesity, diabetes, high blood pressure, high cholesterol, or smoking are associated with an increased risk of events such as myocardial infarction, stroke, or peripheral artery disease. Lifestyle and dietary measures, as well as pharmacological treatments, can help correct these risk factors.

However, several studies have shown that even with optimal treatment, individuals at high risk still face a residual cardiovascular risk. This phenomenon is primarily attributed to the development of vascular lesions, meaning damage within the blood vessels. These lesions are largely due to inflammation, an activated immune state that is more pronounced in overweight individuals and significantly contributes to vascular damage, potentially shortening the lifespan of those with cardiovascular disease.

Although anti-inflammatory therapies have proven effective in reducing this risk, they may interfere with tissue repair and the immune system. For this reason, it is essential to identify strategies that promote the resolution of inflammation without compromising these vital processes.

Specialized pro-resolving mediators (SPMs) are compounds derived from omega-3 and omega-6 polyunsaturated fatty acids, which are naturally found in various foods such as fish. These mediators help limit the infiltration of inflammatory cells and initiate the repair of damaged tissues. This type of dietary supplement is already available over the counter, but its health benefits have not been extensively studied. Experimental animal studies have shown that restoring inflammation resolution through SPMs can prevent-or even reverse-cardiovascular damage and inflammation by directly acting on vascular cells and modulating the immune system. However, human data on the role of SPMs and inflammation resolution in vascular disease remain very limited.

The investigators hypothesize that in individuals at high cardiovascular risk (due to obesity and hypertension), increasing circulating levels of SPMs through oral supplementation (as a dietary supplement) would improve vascular function, metabolic profile, and inflammatory and immune cell responses. In doing so, this may help reduce the residual risk of cardiovascular disease.

The objective of this research is to assess whether a supplement enriched with SPMs can facilitate the resolution of inflammation, which is essential for restoring vascular function and thereby supporting the body's natural tissue repair mechanisms.

To address the research question, the study plans to include 50 individuals with obesity and hypertension, all presenting a high cardiovascular risk, recruited from healthcare facilities located in France.

This research is publicly funded by the French National Research Agency (Agence Nationale de la Recherche) through the European research project RESPIN-VAR, co-funded by ERA4Health and the European Union.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years,.
* Hypertension controlled under pharmacological or non-pharmacological treatment, defined as office BP< 140/90 mmHg at the Inclusion visit,
* BMI > 30 kg/m²,
* Stable antihypertensive treatment one month before inclusion (V1),
* Signed informed consent,
* Social security affiliation.

Exclusion Criteria:

* Secondary hypertension on the basis of medical history,
* History of stroke on the basis of medical history,
* Myocardial infarction on the basis of medical history,
* Severe hepatic insufficiency on the basis of medical history,
* Chronic kidney disease (DFG < 30 ml/min 1.73 according to MDRD method),
* Pregnancy or breast feeding,
* Regular treatment with NO-donors or phosphodiesterase inhibitors,
* Inability to comply with protocol requirements,
* Patient under tutorship or / guardianship or/ safeguard of justice, and incapable to give informed consent,
* Patient on AME (state medical aid),
* Participation in another interventional study involving human participants ,
* Allergy to the ultrasound gel,
* Hypersensitivity , allergy, or idiosyncratic reaction to omega-3 acids, fish or soya allergies.
* Chronic inflammatory diseases, on the basis of medical history,
* Chronic anti-inflammatory treatment administered within the past month preceding the Inclusion visit,
* Any supplementation with omega-3 or omega-6 polyunsaturated fatty acids within the past month,
* Life expectancy less than one year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Flow-mediated dilation (FMD) | FMD will be measured at Week 0 (baseline), Week 12 (after a first administration period of 12 weeks ± 2 days) , Week 14 (after a wash-out period of 2 weeks ± 2 days), Week 26 (after a second administration period of 12 weeks ± 2 days)
  Conduit-artery endothelial function measured by flow-mediated dilation (FMD) after 12 week-intervention with oral SPM supplementation or placebo.

SECONDARY OUTCOMES:
Shear rate area under the curve (SR-AUC) | These parameters will be measured at Week 0 (baseline), Week 12 (after a first administration period of 12 weeks ± 2 days) , Week 14 (after a wash-out period of 2 weeks ± 2 days), Week 26 (after a second administration period of 12 weeks ± 2 days)
  SR-AUC measured as the integral of brachial artery shear rate (flow velocity/diameter*0,8) following post-ischemic reactive hyperemia induced by 5-min forearm cuff occlusion during FMD test
Difference after 12 -week- intervention with oral SPM supplementation or placebo in arterial stiffness | These parameters will be measured at Week 0 (baseline), Week 12 (after a first administration period of 12 weeks ± 2 days) , Week 14 (after a wash-out period of 2 weeks ± 2 days), Week 26 (after a second administration period of 12 weeks ± 2 days)
  Arterial stiffness measured by cfPWV, office brachial and central BP and central hemodynamics measured by Sphygmocor CVMS.
Change from initiation to the end of the 12 -week- intervention in endothelial injury | These parameters will be measured at Week 0 (baseline), Week 12, Week 14, Week 26.
  This outcome assesses endothelial injury by measuring a panel of biological markers that together reflect vascular endothelial function and inflammatory status. The selecting markers includes: panel of 15 markers including sICAM, sVCAM, eSelectin, vWF, based on ELISA (in house assay), electrochemiluminescence (V-PLEX, MesoScale Discoveries) and LuminexTM technologies.) and inflammatory cytokines (16 different cytokines including CRP, SAA, IL-6, IL-8, TNF-a)
Change from initiation to the end of the 12 -week- intervention immune cell profile | These parameters will be measured at Week 0, Week12, Week14, Week26
  A panel of 12 soluble immune checkpoints as potential novel actors in cardiovascular disease will be quantified including sCD25 (IL-2Ra), s4-1BB, sCD27, sCD86 (B7.2), TGF-β1 (free active form), sCTLA-4, and sGalectin-9, among others. PBMCs will be assayed for their activation capabilities by means of multiparametric intracellular spectral flow cytometry in the presence of a polyclonal stimulation.
Insulin sensitivity | These parameters will be measured at Week 0, Week12, Week14, Week26
  Insulin sensitivity will be assessed using the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), calculated from fasting glucose and insulin levels. This outcome evaluates metabolic response to the intervention.
Change in Body Fat Mass | These parameters will be measured at Week 0, Week12, Week14, Week26
  Body fat mass will be measured using a validated smart scale based on bioelectrical impedance. This outcome assesses changes in body composition during the intervention period.
Change in Lipid profile | These parameters will be measured at Week 0, Week12, Week14, Week26
  Serum total cholesterol, HDL cholesterol, and triglycerides concentration will be measured as a marker of lipid metabolism.
Safety assessement by Liver function markers | These parameters will be measured at Week 0, Week12, Week14, Week26
  Description : Liver function markers are AST, ALT, gammaGT
Safety assessement by Renal function markers | These parameters will be measured at Week 0, Week12, Week14, Week26
  Renal function will be evaluated through a composite of serum creatinine, serum uric acid, and urinalysis parameters (albuminuria/creatinuria ratio).
Safety assessement by Coagulation markers | These parameters will be measured at Week 0, Week12, Week14, Week26
  Coagulation function will be evaluated through a composite of prothrombin time and activated partial thromboplastin time.
SPM levels | These parameters will be measured at Week 0, Week12, Week14, Week26
  SPM levels
Questionnaires about perceptions and expectations about oral supplements for cardiovascular disease prevention | Week 0 and Week 26
  Change in Perceptions and Expectations Regarding Oral Supplements for Cardiovascular Disease Prevention
  Participants will complete a questionnaire assessing their perceptions and expectations about the use of oral supplements forcardiovascular disease prevention.
Health Literacy Questionnaire | Week 26
  Participants health literacy will be evaluated at the end of the intervention using a validated health literacy questionnaire. The objective is to assess their ability to access, understand, and use health-related information for decision-making.
Questionnaire about vascular ageing awareness | Week 26
  Questionnaire about vascular ageing awareness

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Maria BRUNO, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Pharmacologie - UF Pharmacologie Clinique, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision. Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).